CLINICAL TRIAL: NCT00659529
Title: The Role of Phosphodiesterase Inhibitors in CF Lung Disease
Brief Title: Safety and Efficacy of Sildenafil in Cystic Fibrosis (CF) Lung Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Jennifer Taylor-Cousar, Principal Investigator, National Jewish Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 851R14-8510M3
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Results first posted 2014-05-02 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; inflammation; pH; EBC; sputum biomarkers; phosphodiesterase inhibitors
MeSH Terms: conditions — Cystic Fibrosis; Inflammation | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All subjects will receive oral sildenafil three times per day during the study. Study endpoints will be measured before the treatment period and at the end of the treatment period.
  Interventions: Drug: sildenafil

INTERVENTIONS:
Drug: sildenafil — Sildenafil will be given 20mg po tid for 1 week, and then will be give 40mg po tid for 5 weeks.
  Other Names: Revatio

SUMMARY:
The purpose of this study is to determine whether sildenafil can decrease inflammation in CF lung disease.

DETAILED DESCRIPTION:
This study is an open-label study that examines the use of sildenafil (Revatio) in clinically stable patients with mild to moderate CF lung disease. The length of participation for each subject will be approximately 10 weeks, and will consist of a screening visit, a study visit for initiation of study drug if subject qualifies, interim visits to escalate drug dose, obtain drug levels, review concomitant medications and assess side effects, a visit at the end of the therapy period (to reassess inflammatory markers, laboratory studies and side effects,) and a follow-up assessment 2 weeks after subject completion.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF based on the following criteria:

  * Positive sweat chloride ≥60mEq/liter (by pilocarpine iontophoresis) and/or
  * Genotype with two identifiable mutations consistent with CF, and accompanied by one or more clinical features consistent with the CF phenotype
* Male or female patients ≥ 12 years of age
* FEV1 ≥ 50% predicted (Knudson) 31
* Clinically stable without evidence of acute upper or lower respiratory tract infection or current pulmonary exacerbation within the 14 days prior to the screening visit
* Ability to reproducibly perform spirometry (according to ATS criteria)
* Ability to produce at least 1mL of sputum spontaneously, or be willing to undergo sputum induction
* Ability to understand and sign a written informed consent or assent and comply with the requirements of the study
* Chronic bacterial colonization (3 documented positive cultures in the prior 2 years of which at least one was obtained in the 3 months prior to randomization)

Exclusion Criteria:

* History of hypersensitivity to sildenafil
* Use of an investigational agent within the 4-week period prior to Visit 1 (Day 0)
* Breastfeeding, pregnant, or verbal expression of unwillingness to practice an acceptable birth control method (abstinence, hormonal or barrier methods, partner sterilization or intrauterine device) during participation in the study
* Daily use of systemic corticosteroids and/or NSAIDs within 4 weeks of the study or as needed use within 72 hours prior to the screening visit
* History of significant hepatic (SGOT or SGPT > 3 times the upper limit of normal at screening, documented biliary cirrhosis, or portal hypertension), cardiovascular (history of aortic stenosis, coronary artery disease, pulmonary hypertension with right ventricular systolic pressure >55 mmHg or life-threatening arrhythmia), neurological (history of stroke), hematologic (history of bleeding diathesis), ophthalmologic (history of retinal impairment or non-arteritic ischemic optic neuritis) or renal impairment (creatinine >1.8 mg/dL.)
* Inability to swallow pills
* Previous lung transplantation
* Use of concomitant nitrates, α-blocker, or Ca channel blocker
* Use of concomitant medications known to be potent inhibitors of CYP3A4 (e.g. ketoconazole, itraconazole, ritonavir, clarithromycin, erythromycin, rifampin)
* Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the subject or the quality of the data
* Weight less than 40 kg
* History of sputum or throat swab culture yielding Burkholderia cepacia within 2 years of screening
* Resting room air oxygen saturation <93%
* History of migraines

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Taylor-Cousar, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poschet JF, Timmins GS, Taylor-Cousar JL, Ornatowski W, Fazio J, Perkett E, Wilson KR, Yu HD, de Jonge HR, Deretic V. Pharmacological modulation of cGMP levels by phosphodiesterase 5 inhibitors as a therapeutic strategy for treatment of respiratory pathology in cystic fibrosis. Am J Physiol Lung Cell Mol Physiol. 2007 Sep;293(3):L712-9. doi: 10.1152/ajplung.00314.2006. Epub 2007 Jun 22. PMID 17586695
- [Derived] Taylor-Cousar JL, Wiley C, Felton LA, St Clair C, Jones M, Curran-Everett D, Poch K, Nichols DP, Solomon GM, Saavedra MT, Accurso FJ, Nick JA. Pharmacokinetics and tolerability of oral sildenafil in adults with cystic fibrosis lung disease. J Cyst Fibros. 2015 Mar;14(2):228-36. doi: 10.1016/j.jcf.2014.10.006. Epub 2014 Nov 13. PMID 25466700

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label (All Subjects): All subjects will receive oral sildenafil three times per day during the study. Study endpoints will be measured before the treatment period and at the end of the treatment period.
  sildenafil: Sildenafil will be given 20mg po tid for 1 week, and then will be give 40mg po tid for 5 weeks.
Period: Overall Study
Arm/Group | Open-label (All Subjects)
Started | 36 (There were 9 screen failures (subjects who did not meet inclusion/exclusion criteria))
Received at Least One Dose of Study Drug | 27 (Received at least one dose of study drug)
Completed | 20 (4 patients withdrew as a result of side effects. 3 subjects were withdrawn by the investigator.)
Not Completed | 16
Not completed — Withdrawal by Subject | 4
Not completed — Protocol Violation | 3
Not completed — Screen failure | 9

BASELINE CHARACTERISTICS:
Population: All patiens who received at least one dose of study drug.
Arm/Group | Open-label (All Subjects)
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.7 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 11
FEV1% predicted [Mean (Standard Deviation); unit: % predicted] | 77.5 (19.6)

OUTCOME MEASURES:

1. Primary Outcome: Sputum Elastase
Time Frame: Pre/post therapy
Population: Subjects who completed 6 weeks of sildenafil and had available data for pre/post 6 weeks of sildenafil were analyzed. One subject presented to the final study visit with 1 week of previously unreported symptoms consistent with pulmonary exacerbation, and therefore, efficacy data was not analyzed on that subject as pre-specified in the protocol.
Measure: Mean (95% Confidence Interval); unit: micrograms/mL
Arm/Group | Open-label (All Subjects)
Number analyzed (Participants) | 18
micrograms/mL | -57 [-119 to -18]

2. Secondary Outcome: Exhaled Breath Condensate pH
Time Frame: Pre/post therapy
Reporting Status: Not Posted

3. Secondary Outcome: CFQ-R
Time Frame: Pre/post therapy
Reporting Status: Not Posted

4. Secondary Outcome: Serum Sildenafil Levels
Time Frame: Pre/during therapy
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Open-label (All Subjects)
Serious Adverse Events (participants affected / at risk) | 2/27
Other Adverse Events (participants affected / at risk) | 24/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label (All Subjects) (N=27)
CF pulmonary exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Distal Intestinal Obstruction Syndrome (Gastrointestinal disorders) | 1 (1) — Not related to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label (All Subjects) (N=27)
headache (Nervous system disorders) | 6
rhinorhhea/congestion (Respiratory, thoracic and mediastinal disorders) | 9
Sore throat/throat clearing (General disorders) | 6
Increased cough (Respiratory, thoracic and mediastinal disorders) | 6
Flushing (General disorders) | 5
dyspepsia (Gastrointestinal disorders) | 4
myalgia (Musculoskeletal and connective tissue disorders) | 4
Increased/thicker sputum (Respiratory, thoracic and mediastinal disorders) | 4
Insomnia (General disorders) | 3
Chest tigntness/congestion (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No